CLINICAL TRIAL: NCT00873288
Title: Activating Collaborative CIS Support Via Targeted Provider Mailing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bonnie Spring, Director, Center for Behavior and Health, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CDR0000626557; P30CA060553 (NIH); NU-1719-007 (Other: Northwestern University); R21CA126450 (NIH)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Precancerous Condition
Keywords: cervical intraepithelial neoplasia; atypical squamous cells of undetermined significance; high-grade squamous intraepithelial lesion; low-grade squamous intraepithelial lesion
MeSH Terms: conditions — Precancerous Conditions; Uterine Cervical Dysplasia; Atypical Squamous Cells of the Cervix; Squamous Intraepithelial Lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care mailing intervention (Active Comparator): routine colposcopy reminder letter mailed
  Interventions: Other: Usual care mailing intervention
- CIS support mailing intervention (Experimental): Mailed reminder plus provider recommendation to call CIS and sample questions to ask
  Interventions: Other: CIS support mailing intervention

INTERVENTIONS:
Other: Usual care mailing intervention — routine colposcopy reminder letter
  Arms: Usual Care mailing intervention
Other: CIS support mailing intervention — Mailed reminder plus provider recommendation to call CIS and sample questions to ask
  Arms: CIS support mailing intervention

SUMMARY:
RATIONALE: Receiving a reminder letter from their doctor with questions to ask the Cancer Information Service may be more effective than a standard reminder letter in helping patients who have had an abnormal Pap test keep their follow-up colposcopy appointment.

PURPOSE: This randomized clinical trial is studying a personalized letter with Cancer Information Service support to see how well it works compared with a standard reminder letter in women scheduled for colposcopy after an abnormal Pap test.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of a usual care mailing intervention vs a Cancer Information Service (CIS) support mailing intervention on the likelihood that women with an abnormal Pap test will keep their medical follow-up appointments and be satisfied with how they talk to their provider.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 intervention arms.

* Arm I (Usual-care mailing intervention): Patients receive a generic letter reminding them of their follow-up colposcopy appointment.
* Arm II (Cancer Information Service [CIS] support mailing intervention): Patients receive a targeted letter reminding them of their follow-up colposcopy appointment, asking them or someone they designate to call the CIS, and suggesting some questions to ask the CIS about colposcopies and Pap tests.

At their follow-up appointments, all patients undergo an exit interview to compare patient satisfaction between the 2 interventions. Patients in arm II also answer questions about their CIS experience, and if the intervention made their follow-up visit less difficult.

ELIGIBILITY:
Inclusion criteria:

DISEASE CHARACTERISTICS:

* Received an abnormal Pap test result
* Scheduled for a colposcopy within 6 months of their Pap test at either the Erie Family Health Center or the Prentice Ambulatory Clinic

PATIENT CHARACTERISTICS:

* Female
* Able to communicate in either English or Spanish
* Clinic staff will review patient charts to determine eligibility

PRIOR CONCURRENT THERAPY:

* Not specified

Exclusion criteria:

* <18 years
* unable to communicate in English or Spanish
* no address to which a letter can be mailed

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Erie Family Health Center, Chicago, Illinois

REFERENCES:
- [Background] Cofta-Woerpel L, Randhawa V, McFadden HG, Fought A, Bullard E, Spring B. ACCISS study rationale and design: activating collaborative cancer information service support for cervical cancer screening. BMC Public Health. 2009 Dec 2;9:444. doi: 10.1186/1471-2458-9-444. PMID 19951443
- [Background] Simon MA, Cofta-Woerpel L, Randhawa V, John P, Makoul G, Spring B. Using the word 'cancer' in communication about an abnormal Pap test: finding common ground with patient-provider communication. Patient Educ Couns. 2010 Oct;81(1):106-12. doi: 10.1016/j.pec.2009.11.022. Epub 2010 Jan 8. PMID 20060255

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Started | 127 | 127
Completed | 127 | 127
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention | Total
Number analyzed (Participants) | 127 | 127 | 254
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 127 | 254
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (9.1) | 27.8 (9.3) | 27.95 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 127 | 254
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 127 | 254

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction in the 2 Interventions
Description: Patient satisfaction with provider-patient communication was assessed via administration of the Consumer Assessment of Health Plans Study (CAHPS) satisfaction questionnaire which rates satisfaction on a 1 to 3 scale. Scores are added together, with minimum score being 4 and the maximum score being 12, with a higher score indicating greater satisfaction.
Time Frame: within 6 months of PAP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Number analyzed (Participants) | 127 | 127
score on a scale | 11.79 (.563) | 11.68 (.912)
Statistical Analysis 1: Comparison: Usual Care Mailing Intervention vs CIS Support Mailing Intervention; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Primary Outcome: CIS Experience of Patients in Arm II and the Effect of the Intervention on Their Follow-up Colposcopy
Time Frame: within 6 months of PAP
Population: The apparatus that Boeing built to identify which CIS callers were from the study did not function correctly. Therefore, we could not determine whether participants called CIS or not.
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Attendance at a Follow-up Colposcopy Appointment Within 6 Months of Their Pap Test
Time Frame: within 6 months of PAP
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Number analyzed (Participants) | 127 | 127
Participants | 107 | 102
Statistical Analysis 1: Comparison: Usual Care Mailing Intervention vs CIS Support Mailing Intervention; Test type: Superiority; p = 0.207, Chi-squared; The Pearson Chi-squared value = 1.590

4. Secondary Outcome: Latency Between the Pap Test and the Colposcopy Appointment
Time Frame: within 6 months of PAP
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Number analyzed (Participants) | 127 | 127
days | 39.5 [29 to 55] | 42.5 [30 to 66]
Statistical Analysis 1: Comparison: Usual Care Mailing Intervention vs CIS Support Mailing Intervention; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

5. Secondary Outcome: Number of CIS Callers Who Provided the Specific Codes Listed in the Intervention Letter
Time Frame: WITHIN 6 MONTHS OF PAP
Population: as for outcome 2
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Usual Care Mailing Intervention | CIS Support Mailing Intervention
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/127
Other Adverse Events (participants affected / at risk) | 0/127 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No